CLINICAL TRIAL: NCT04273867
Title: Assessing Health Related Quality of Life in Hypersensitivity Pneumonitis
Acronym: CHP-HRQOL
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pulmonary Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-05020233
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hypersensitivity Pneumonitis; Chronic Hypersensitivity Pneumonitis; Interstitial Lung Disease; Extrinsic Allergic Alveolitis; Health-related Quality of Life
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Hypersensitivity Pneumonitis Patients
  Interventions: Other: Chronic Hypersensitivity Pneumonitis Health Related Quality of Life Survey Instrument

INTERVENTIONS:
Other: Chronic Hypersensitivity Pneumonitis Health Related Quality of Life Survey Instrument — This survey has been developed and revised from prior qualitative research with CHP patients and will be used to better evaluate disease status and quality of life with CHP.

SUMMARY:
The objective of this study is to administer and validate a disease specific health related quality of life (HRQOL) survey for patients with Chronic Hypersensitivity Pneumonitis (CHP).

DETAILED DESCRIPTION:
The objective of this study is to administer and validate a disease-specific health related quality of life (HRQOL) survey for patients with Chronic Hypersensitivity Pneumonitis (CHP). The survey items have been developed and revised from prior qualitative research with CHP patients. Potential participants will be recruited from WCMC, the Pulmonary Fibrosis Foundation (PFF) Registry and outside physician referral for the study. Participants will be asked to sign informed consent. At the initial visit participants will be asked to complete the survey and two additional PROs needed for concurrent validity testing. Participants will then be asked to complete the HRQOL survey under study a second time 2 weeks after the initial visit for test-re-test reliability testing. Pulmonary function testing and six minute walk test results will be collected. Pertinent demographic and clinical information will be collected from the patients and their medical records or registry data (if a PFF Registry participant). All information will be entered into a REDCap database for secure data management and storage. Psychometric testing will be performed on the overall survey instrument and the individual items in order to test validity and reliability. The goal is that the survey developed will be a reliable and valid measurement tool for use in both clinical practice and research settings.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Understand and sign the informed consent document
3. Documented diagnosis of HP made and confirmed at an ILD center via expert consensus or in multidisciplinary discussion

   a. Diagnosis based upon a minimum of a medical history, physical examination, pulmonary function testing, and computerized tomography (CT) scan. Pathology will be reviewed if available but is not required.
4. HP must be the primary pulmonary disease
5. Anticipated ability to complete follow up survey within 2 weeks of initial survey completion
6. Participants recruited from the PFF registry must have agreed to be contacted for ancillary research studies.

Exclusion Criteria:

1. Non-English Speaking (Patient must be able to speak and read English fluently but it does not have to be their primary language)
2. Inability to complete questionnaire due to cognitive impairment
3. Patients who have not been seen by or communicated with their provider in over 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in many ways including i2b2 search in Electronic Medical Record (EMR) (EPIC) for patients with diagnosis code for Hypersensitivity Pneumonitis, or Extrinsic Allergic Alveolitis (ICD 10: J67.9), weekly review of scheduled office visits in the EMR for patients with diagnosis of Hypersensitivity Pneumonitis, multi-disciplinary conference discussions of patients with a diagnosis of Chronic Hypersensitivity Pneumonitis, physician Referrals from both WCM and local outside institutions, recruitment flyers, and patient support groups
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Validation of a health-related quality of life instrument for patients with Chronic Hypersensitivity Pneumonitis | Day 0
  The newly developed survey that is being validated consists of 42 items that assess the impact that Hypersensitivity Pneumonitis has on daily life for those who have the disease.
Validation of a health-related quality of life instrument for patients with Chronic Hypersensitivity Pneumonitis by administering the Short Form (SF-12) Survey | Day 0
  This survey will be used to assess the validity of the newly developed health-related quality of life instrument. This survey consists of 12 items. The average score for this survey has been calibrated to 50 with scores below 50 indicating a below average score and scores above 50 indicating an above average score.
Validation of a health-related quality of life instrument for patients with Chronic Hypersensitivity Pneumonitis by administering the King's Brief Interstitial Lung Disease Questionnaire | Day 0
  This survey will be used to assess the validity of the newly developed health-related quality of life instrument. This survey consists of 15 items and is scored from 0-100 with 100 indicating good health.
Change in Health-related Quality of Life Assessment Score | 2 weeks following Day 0
  The newly developed survey will be administered again in 2 weeks following the first assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri I Aronson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No